CLINICAL TRIAL: NCT01365169
Title: "CYCORE: Cyberinfrastructure for Comparative Effectiveness Research - Feasibility Trial"
Brief Title: Association Between Health Care Provider (HCP)-Assessed ECOG Performance Status (PS) and Overall Survival, and Objectively Measure of Physical Activity (PA) Levels in Advance-cancer Patients"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010-0955; NCI-2014-02468 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0955 (Other: M D Anderson Cancer Center); R01CA243554 (NIH); RC2CA148263 (NIH); R01CA177996 (NIH)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Malignant Head and Neck Neoplasm; Malignant Neoplasm; Metastatic Malignant Neoplasm in the Neck; Metastatic Malignant Neoplasm in the Uterine Cervix; Pancreatic Adenocarcinoma; Pancreatic Neuroendocrine Carcinoma; Recurrent Colorectal Carcinoma; Stage I Colorectal Cancer AJCC v6 and v7; Stage I Hypopharyngeal Carcinoma AJCC v7; Stage I Major Salivary Gland Cancer AJCC v7; Stage I Nasopharyngeal Carcinoma AJCC v7; Stage I Oral Cavity Cancer AJCC v6 and v7; Stage I Oropharyngeal Carcinoma AJCC v6 and v7; Stage II Colorectal Cancer AJCC v7; Stage II Hypopharyngeal Carcinoma AJCC v6 and v7; Stage II Major Salivary Gland Cancer AJCC v7; Stage II Nasopharyngeal Carcinoma AJCC v7; Stage II Oral Cavity Cancer AJCC v6 and v7; Stage II Oropharyngeal Carcinoma AJCC v6 and v7; Stage IIA Colorectal Cancer AJCC v7; Stage IIB Colorectal Cancer AJCC v7; Stage IIC Colorectal Cancer AJCC v7; Stage III Colorectal Cancer AJCC v7; Stage III Hypopharyngeal Carcinoma AJCC v7; Stage III Laryngeal Cancer AJCC v6 and v7; Stage III Major Salivary Gland Cancer AJCC v7; Stage III Nasopharyngeal Carcinoma AJCC v7; Stage III Oral Cavity Cancer AJCC v6 and v7; Stage III Oropharyngeal Carcinoma AJCC v7; Stage IIIA Colorectal Cancer AJCC v7; Stage IIIB Colorectal Cancer AJCC v7; Stage IIIC Colorectal Cancer AJCC v7; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVA Hypopharyngeal Carcinoma AJCC v7; Stage IVA Laryngeal Cancer AJCC v7; Stage IVA Major Salivary Gland Cancer AJCC v7; Stage IVA Nasopharyngeal Carcinoma AJCC v7; Stage IVA Oral Cavity Cancer AJCC v6 and v7; Stage IVA Oropharyngeal Carcinoma AJCC v7; Stage IVB Colorectal Cancer AJCC v7; Stage IVB Hypopharyngeal Carcinoma AJCC v7; Stage IVB Laryngeal Cancer AJCC v7; Stage IVB Major Salivary Gland Cancer AJCC v7; Stage IVB Nasopharyngeal Carcinoma AJCC v7; Stage IVB Oral Cavity Cancer AJCC v6 and v7; Stage IVB Oropharyngeal Carcinoma AJCC v7; Metastatic or Locally Unresectable Solid Tumor
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Somatostatinoma; Colorectal Neoplasms; Hypopharyngeal Neoplasms; Nasopharyngeal Carcinoma; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm I (colorectal cancer patients) (Experimental): (CLOSED TO ACCRUAL AS OF 01/30/14) Patients use two accelerometers, a blood pressure monitor, a heart rate monitor, a GPS device, and a smart phone that prompts patients to electronically answer questions about exercise and health-related symptoms and feelings. The devices are used for 5 consecutive days. After a 2 week period, patients resume use of the devices for an additional 5 days.
  Interventions: Other: Health Telemonitoring; Other: Questionnaire Administration
- Arm II (head and neck cancer patients) (Experimental): (CLOSED TO ACCRUAL AS OF 01/30/14) Patients use two accelerometers, a blood pressure monitor, a weight scale, and a smart phone that prompts patients to electronically answer questions about diet and health-related symptoms. The devices are used for 5 consecutive days. After a 2 week period, patients resume use of the devices for an additional 5 days.
  Interventions: Other: Health Telemonitoring; Other: Questionnaire Administration
- Arm III (head and neck cancer patients) (Experimental): (CLOSED TO ACCRUAL AS OF 01/30/14) Patients use a smart phone that prompts patients to electronically answer questions about diet, health-related symptoms, and swallowing exercises. Patients also take video recordings of their neck while performing swallowing exercises. The device is used for 5 consecutive days. After a 2 week period, patients resume use of the device for an additional 5 days.
  Interventions: Other: Health Telemonitoring; Other: Questionnaire Administration
- Arm IV (cancer survivors that are current/former smokers) (Experimental): (CLOSED TO ACCRUAL AS OF 01/30/14) Patients use a CO monitor and a smart phone that prompts patients to electronically answer questions about smoking. Patients also take video recordings of themselves while exhaling into the CO monitor. The devices are used for 5 consecutive days. After a 2 week period, patients resume use of the devices for an additional 5 days.
  Interventions: Other: Health Telemonitoring; Other: Questionnaire Administration
- PCS (pancreatic surgery patients) (Experimental): Patients receive post-surgical wellness program consisting of physical activity, nutrition counseling, and daily monitoring (physical activity, weight, and self-reported data) for up to 7 months post-op.
  Interventions: Behavioral: Exercise Intervention; Other: Health Telemonitoring; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- TAPS (Technological Approach to Performance Status) (Experimental): Patients use two Physical Activity monitor devices, the wrist-worn device (Fitbit) continuously and the Actigraph during waking hours. Patients use the devices for 7 consecutive days.
  Interventions: Other: Health Telemonitoring

INTERVENTIONS:
Behavioral: Exercise Intervention — Participate in walking and/or strengthening program
  Arms: PCS (pancreatic surgery patients)
Other: Health Telemonitoring — Use accelerometers, blood pressure monitor, heart rate monitor, GPS device, and smart phone
  Arms: Arm I (colorectal cancer patients)
Other: Health Telemonitoring — Use accelerometers, blood pressure monitor, weight scale, and smart phone
  Arms: Arm II (head and neck cancer patients)
Other: Health Telemonitoring — Use smart phone
  Arms: Arm III (head and neck cancer patients)
Other: Health Telemonitoring — Use CO monitor and smart phone
  Arms: Arm IV (cancer survivors that are current/former smokers)
Other: Health Telemonitoring — Use Fitbit, weight scale and iPhone- or web-based app for self-reported data
  Arms: PCS (pancreatic surgery patients)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: PCS (pancreatic surgery patients)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (colorectal cancer patients); Arm II (head and neck cancer patients); Arm III (head and neck cancer patients); Arm IV (cancer survivors that are current/former smokers); PCS (pancreatic surgery patients)
Other: Health Telemonitoring — Use Fitbit and Actigraph
  Arms: TAPS (Technological Approach to Performance Status)

SUMMARY:
The main goal of this phase of the study is to determine if objectively assessed Physical Activity (PA) levels in advanced-cancer patients are associated with health care provider (HCP)-assessed ECOG performance status and overall survival. The purpose is to advance the evidence-base for incorporating objective assessment of Physical Activity (PA) in the context of performance status assessment in advanced cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the feasibility and acceptability in diverse samples of cancer patients of wireless collection and transmission of data for transfer into the open-source cyberinfrastructure (CI) called Cyberinfrastructure for Comparative Effectiveness Research (CYCORE).

OUTLINE: Patients are assigned to 1 of 4 arms.

ARM I (COLORECTAL CANCER PATIENTS) (CLOSED TO ACCRUAL AS OF 01/30/14): Patients use two accelerometers, a blood pressure monitor, a heart rate monitor, a global positioning system (GPS) device, and a smart phone that prompts patients to electronically answer questions about exercise and health-related symptoms and feelings. The devices are used for 5 consecutive days. After a 2 week period, patients resume use of the devices for an additional 5 days.

ARM II (HEAD AND NECK CANCER PATIENTS) (CLOSED TO ACCRUAL AS OF 01/30/14): Patients use two accelerometers, a blood pressure monitor, a weight scale, and a smart phone that prompts patients to electronically answer questions about diet and health-related symptoms. The devices are used for 5 consecutive days. After a 2 week period, patients resume use of the devices for an additional 5 days.

ARM III (HEAD AND NECK CANCER PATIENTS) (CLOSED TO ACCRUAL AS OF 01/30/14): Patients use a smart phone that prompts patients to electronically answer questions about diet, health-related symptoms, and swallowing exercises. Patients also take video recordings of their neck while performing swallowing exercises. The device is used for 5 consecutive days. After a 2 week period, patients resume use of the device for an additional 5 days.

ARM IV (CANCER SURVIVORS THAT ARE CURRENT/FORMER SMOKERS) (CLOSED TO ACCRUAL AS OF 01/30/14): Patients use a carbon monoxide (CO) monitor and a smart phone that prompts patients to electronically answer questions about smoking. Patients also take video recordings of themselves while exhaling into the CO monitor. The devices are used for 5 consecutive days. After a 2 week period, patients resume use of the devices for an additional 5 days.

PANCREATIC CANCER STUDY (PCS): Patients receive post-surgical wellness program consisting of physical activity, nutrition counseling, and daily monitoring (physical activity, weight, and self-reported data) for up to 7 months post-op.

Technological Approach to Performance Status (TAPS) Study: Patients use two Physical Activity monitor devices, the wrist-worn device (Fitbit) continuously and the Actigraph during waking hours. Patients use the devices for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any stage I - IV colorectal cancer or recurrent colorectal cancer (Arm 1)
* Able to speak, read, and write in English (Pre-pilot phase, Arms 1-4)
* Able to provide informed consent (Pre-pilot phase, Arms 1-4, PCS study)
* Lives in the Houston area (Harris county or a contiguous county) (Pre-pilot phase)
* Eastern Cooperative Oncology Group (ECOG) status of 0 - 2, or self-reports being up and about more than 50% of waking hours and able to provide self-care (Arm 1)
* Diagnosis of any of the following cancers: stage 1-4b oropharyngeal, hypopharyngeal, nasopharyngeal, salivary gland or oral cavity; stage 3-4b laryngeal; any unknown primary head and neck cancer with cervical metastasis that will be addressed with treatment to bilateral necks and mucosa; or other head and neck cancers medically approved by one of our Radiation Oncology collaborating medical doctors (MDs) (Arms 2 and 3)
* History of any cancer, other than non-melanoma skin cancer (Arm 4)
* Admitted to being a current smoker or recent quitter upon admission to MD Anderson Cancer Center (MDACC) (Arm 4)
* Has a valid home address and functioning home telephone number (Arm 4)
* Lives in the Houston or surrounding area, or resides in this same area during the time period that coincides with this study (Arms 1-4)
* Patients who will undergo curative pancreatectomy for pancreatic adenocarcinoma, pancreatic neuroendocrine tumors, or pancreatic cysts (malignant or benign) (PCS study)
* Fluent in English (PCS study)
* Must have telephone access and agree to engage with research personnel using telephone (PCS study)
* Diagnosis of a metastatic or locally unresectable solid tumor (TAPS study)
* Fluent in English (TAPS study)
* Age 18 years or older (TAPS study)
* ECOG performance status score between 0-3 (TAPS study)

Exclusion Criteria:

* Major surgery in the past 8 weeks (Arms 1 and 4)
* Self-reports hypertension that is not being monitored by a physician and is not being managed with either medication, observation, or lifestyle change (Pre-pilot phase, Arms 1-3)
* Overt cognitive difficulty demonstrated by not being clearly oriented to time or person or place (Arms 1-4)
* Orthopedic, neurologic, or musculoskeletal disability that would interfere with the functional task of standing on a weight scale (Pre-pilot phase, Arm 2)
* Not currently receiving radiation treatment for a cancer listed in the arm-specific inclusion criteria (Arms 2 and 3)
* Zubrod performance status > 2, or self-reports either not being up and about more than 50% of waking hours or unable to provide self-care (Arms 2 and 3)
* Currently receiving treatment for a cancer other than those listed in the arm-specific inclusion criteria (exception: the study does not exclude those receiving treatment for non-melanoma skin cancer) (Arms 2 and 3)
* History of current oropharyngeal dysphagia unrelated to cancer diagnosis (e.g. dysphagia due to underlying neurogenic disorder) (Arm 3 only)
* Active substance use disorder (diagnosed or strongly suspected) (Arm 4)
* Currently enrolled in protocol 2014-0712 (PCS study)
* No home access to internet (PCS study)
* No home WiFi connection (PCS study)
* During clinician's pre-surgical evaluation, presents with high risk for non-therapeutic resection related to cancer diagnosis (PCS study)
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease (New York Heart Association functional class III or IV) (PCS study)
* Recent fracture or acute musculoskeletal injury that precludes the ability to fully bear weight on all 4 limbs in order to participate in an exercise intervention (PCS study)
* Poorly-controlled pain with a self-reported pain score of 7/10 at the time of enrollment (PCS study)
* Myopathic or rheumatologic disease that impacts physical function (PCS study)
* Has a pacemaker or other internal medical device, or reports being pregnant (PCS study)
* Currently enrolled in protocol 2017-0198 (PCS study)
* Demonstration of overt cognitive difficulty as demonstrated by not being clearly oriented to time or person or place (TAPS study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2011-05-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Study completion (defined as completing the final assessment) | Up to 7 months after baseline
Physical Activity (PA) Assessment | Up to 7 days
  PA will be measured by two different devices, (1) a consumer-grade wrist-worn device that collects continuous PA data (Fitbit), and (2) a research-grade, hip-worn accelerometer (Actigraph)
ECOG Performance Status | Up to 2 weeks
  Eastern Cooperation Oncology Group (ECOG) is a 6-point performance status scale used to assess performance using PA as a key indicator (e.g., 0 = fully active, 2 = up and about more than 50% of walking hours, 5 = dead) Performance status will be assessed per usual clinical practice and will be recorded in the medical record.

SECONDARY OUTCOMES:
Correlation between PA data from the Actigraph and Fitbit | Up to 7 days
  Association between PA measured using a Fitbit and PA measured using Actigraph
Correlation between patients' ECOG performance status scores and PA data | Up to 7 days
  Association between performance status (PS) assesses by the patient's medical oncologist, and PA data
Correlation between PA data and Overall Survivor (OS) | Up to 7 days
  Association between Physical Activity (PA) data and the Overall Survivor (OS) rate
Accrual of Diverse Sample of Cancer-Patients | Up to 2 weeks
Retention of using home-based health monitor devices (e.g. Fitbit, Actigraph, CO monitor, weight scales) among participants. | Up to 2 weeks
Acceptability of using home-based health monitor devices (e.g. Fitbit, Actigraph, CO monitor, weight scales) among participants. | Up to 2 weeks
Participants ability to activate, set-up, and use the home-based health monitor devices (e.g. Fitbit, Actigraph, CO monitor, weight scales). | Up to 2 weeks
Adherence to procedures for home-based health monitor devices activation (e.g. Fitbit, Actigraph, CO monitor, weight scales) self-monitoring (e.g. PA, weight), and self-reported data capture by the devices. | Up to 2 weeks
Successful upload of data from the home-based health monitor devices to the Cyberinfrastructure for Comparative effectiveness Research (CYCORE) for future analysis. | Up to 2 weeks
CYCORE Data availability for clinicians and researchers in order to be able to daily monitor patients using home-based health monitor devices (e.g. Fitbit, Actigraph, CO monitor, weight scales). | Up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Peterson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org